CLINICAL TRIAL: NCT01838317
Title: A Phase II Study of Pioglitazone for Patients With Cancer of the Pancreas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Muhammad Beg, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 072012-036
Record Dates: First submitted 2013-04-16; First posted 2013-04-24 (Estimated); Results first posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Cancer of the Pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pioglitazone & Chemotherapy in Patients without Diabetes (Experimental)
  Interventions: Drug: Pioglitazone
- Pioglitazone & Chemotherapy in Patients with Diabetes (Experimental)
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone

SUMMARY:
This study is being done to determine whether or not addition of the oral medication, pioglitazone to standard chemotherapy, results in improvement of blood tests that measure the body's ability to utilize sugar (glucose and insulin metabolism). In addition the investigators want to determine whether or not treatment with pioglitazone results in (1) improvement in the size of the tumor, (2) weight gain, (3) improved ability to function during the day and (4) quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Histologically proven adenocarcinoma of the pancreas
* Radiologically measurable disease
* ECOG functional status 0-2

Exclusion Criteria:

* Prior radiation therapy for pancreatic cancer If chemotherapy is planned, new chemotherapy regimen should have started more than 14 days prior to enrollment
* Surgery or radiation planned within 8 weeks of starting therapy
* Prior exposure to Thiazolidinedione (TZD) therapy in the past 12 months
* Hypersensitivity of TZD
* New York heart association class III/IV heart failure.
* Known HIV positive
* Pregnant or lactating women
* History of, or active bladder cancer
* Inadequate hepatic function documented within 14 days of enrollment
* Total bilirubin level > 1.5 x ULN
* AST and ALT > 2.5 x ULN, unless there are liver metastases in which case AST and ALT or > 5 x ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-05; Primary Completion 2017-09-20 (Actual); Study Completion 2017-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Beg, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Pioglitazone and Chemotherapy Without Diabetes; Pioglitazone and Chemotherapy - With Diabetes: 45 mg Pioglitazone daily for 8 weeks and continued chemotherapy throughout 10 week study period.
Period: Overall Study
Arm/Group | Pioglitazone and Chemotherapy Without Diabetes | Pioglitazone and Chemotherapy - With Diabetes
Started | 9 | 5
Completed | 9 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pioglitazone and Chemotherapy in Patients Without Diabetes; Pioglitazone and Chemotherapy in Patients With Diabetes: 45 mg Pioglitazone daily for 8 weeks and continued chemotherapy throughout 10 week study period.
- Total: Total of all reporting groups
Arm/Group | Pioglitazone and Chemotherapy in Patients Without Diabetes | Pioglitazone and Chemotherapy in Patients With Diabetes | Total
Number analyzed (Participants) | 9 | 5 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: All Participants received the same treatment. However, results were analyzed separating those individuals with and without diabetes.
  years
    Pioglitazone and Chemotherapy - Without Diabetes | 58.26 (8.52) | 64.84 (8.87) | 61.55 (8.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 3 | 2 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Adiponectin Level
Description: We will obtain serum levels of adiponectin at baseline and after 8 weeks of treatment with pioglitazone.
Time Frame: Baseline and 8 weeks of treatment with pioglitazone
Measure: Mean (Standard Deviation); unit: μg/ml
Arm/Group | Pioglitazone and Chemotherapy Without Diabetes | Pioglitazone and Chemotherapy - With Diabetes
Number analyzed (Participants) | 9 | 5
μg/ml | 34.47 (27.42) | 29.77 (12.06)

2. Primary Outcome: Change in Standard Glucose Tolerance Test
Description: We will perform the area under the oral glucose tolerance test at baseline and after 8 weeks of treatment with pioglitazone.
Time Frame: Baseline to 120 minutes post glucose bolus
Population: The data was not collected for standard glucose tolerance test.
Arm/Group | Pioglitazone and Chemotherapy Without Diabetes | Pioglitazone and Chemotherapy - With Diabetes
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Glucose to Insulin Ratio
Description: Glucose to insulin ratio will be measured by taking the ratio of fasting level of serum glucose and insulin.
  We will obtain serum levels of fasting glucose and insulin every four weeks in all patients receiving pioglitazone
Time Frame: Every 4 weeks while receiving treatment, up to 8 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Pioglitazone and Chemotherapy Without Diabetes | Pioglitazone and Chemotherapy - With Diabetes
Number analyzed (Participants) | 9 | 5
ratio | 0.81 (13.54) | -6.23 (0.08)

4. Secondary Outcome: Change in Weight
Description: To describe changes in weight in patients with pancreas cancer receiving pioglitazone.
Time Frame: Baseline and every two weeks for 10 weeks, change between baseline and week 10 reported.
Population: There was only 1 patient with data for "with Diabetes" arm, thus Standard Deviation for outcome is 0 for that arm
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Pioglitazone and Chemotherapy Without Diabetes | Pioglitazone and Chemotherapy - With Diabetes
Number analyzed (Participants) | 9 | 1
kg | 2.57 (3.98) | -4.01 (0)

5. Secondary Outcome: Number of Patients With Objective Response
Description: Objective response is the proportion of patients with confirmed complete response (CR) or confirmed partial response (PR) according to the Response Evaluation Criteria in Solid Tumors (RECIST).
Time Frame: 8 weeks of treatment with pioglitazone
Population: Tumor assessment not collected. Data was not collected .
Arm/Group | Pioglitazone and Chemotherapy Without Diabetes | Pioglitazone and Chemotherapy - With Diabetes
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Patients' Performance Status by the Eastern Oncology Cooperative Group (ECOG) Scale of Performance Status
Description: The ECOG Scale of Performance Status measures patients' performance status. Possible grades range from 0 to 5, with lower grade indicating a better performance status.
Time Frame: Baseline and 8 weeks of treatment with pioglitazone
Population: Data was not collected.
Arm/Group | Pioglitazone and Chemotherapy Without Diabetes | Pioglitazone and Chemotherapy - With Diabetes
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Quality of Life by the FACT-Hep Scale
Description: The FACT-Hep Scale (version 4) measures quality of life, It consists of five subscales: (1) physical well-being (PWB); (2) social and family well-being (SFWB); (3) emotional well-being (EWB); (4) functional well-being (FWB); and the hepatobiliary cancer subscale (HepCS). Possible scores range from 0 to 180, with lower scores indicating a better quality of life
Time Frame: Baseline and 8 weeks of treatment with pioglitazone
Population: Data was not collected
Arm/Group | Pioglitazone and Chemotherapy Without Diabetes | Pioglitazone and Chemotherapy - With Diabetes
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in Pancreatic Intratumor Fat
Description: Change in pancreatic intratumor fat will be measured by MRI
Time Frame: Baseline and 8 weeks of treatment with pioglitazone
Population: Data was not collected.
Arm/Group | Pioglitazone and Chemotherapy Without Diabetes | Pioglitazone and Chemotherapy - With Diabetes
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change in Body Fast Distribution
Description: Change in body fast distribution will be measured by MRI
Time Frame: Baseline and 8 weeks of treatment with pioglitazone
Population: This data was not collected as the number of cases with pre and post scans who were with and without DM (Diabetes Mellitus) was too small.
Arm/Group | Pioglitazone and Chemotherapy Without Diabetes | Pioglitazone and Chemotherapy - With Diabetes
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Changes in Serum and MRI End Points
Description: Compare changes in serum and MRI end points between pioglitazone
Time Frame: Baseline and 8 weeks of treatment with pioglitazone
Population: as for outcome 9
Arm/Group | Pioglitazone and Chemotherapy Without Diabetes | Pioglitazone and Chemotherapy - With Diabetes
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 years, 4 months
Arm/Group | Pioglitazone and Chemotherapy Without Diabetes | Pioglitazone and Chemotherapy - With Diabetes
All-Cause Mortality (participants affected / at risk) | 9/9 | 5/5
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/5
Other Adverse Events (participants affected / at risk) | 0/9 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-25): https://cdn.clinicaltrials.gov/large-docs/17/NCT01838317/Prot_SAP_000.pdf